CLINICAL TRIAL: NCT04645589
Title: Evaluating the Safety of Myfortic (Mycophenolate Sodium) in Patients With Lupus Nephritis: a 12 Month, Single-arm, Observational Study in Taiwan Population
Brief Title: Evaluating the Safety of Myfortic (Mycophenolate Sodium) in Patients With Lupus Nephritis
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CERL080ATW12
Record Dates: First submitted 2020-11-23; First posted 2020-11-27 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; LN; Myfortic; Mycophenolate sodium
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myfortic: Oral administration
  Interventions: Drug: Myfortic

INTERVENTIONS:
Drug: Myfortic — There is no treatment allocation. Patients administered Myfortic by prescription that have started before inclusion of the patient into the study will be enrolled.
  Other Names: Mycophenolate sodium

SUMMARY:
This is an open-label, prospective, single-arm, observational study in patients with Lupus nephritis (LN) who newly (i.e.,for the first time) received treatment of Enteric-coated Mycophenolate Sodium (EC-MPS).

DETAILED DESCRIPTION:
This is an observational study. Patients will be treated and followed according to routine medical practice in terms of visit frequency and type of assessment performed. Only endpoint related data will be collected as part of the study. Patient demographic information, disease characteristics, treatments and laboratory data will be collected retrospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 20 years and ≤ 75 years at screening.
2. Patients with written informed consent form.
3. Male or female diagnosed with SLE.
4. Confirmed diagnosis of LN by physician. Diagnosis of LN is defined as:

   a. Kidney biopsy within 1 year, with histological diagnosis of LN (class III/IV/V)
5. Laboratory evidence of active nephritis: spot UPCR>0.5, and/or proteinuria > 0.5 g/24 hours, and/or greater than 3+ by dipstick, and/or cellular casts.
6. Patients with LN who received EC-MPS for the first time. The patients who switched from other treatment and treatment naive patients (did not received any treatment before) can be included in this study.
7. Women of childbearing potential must use effective contraception before beginning EC MPS therapy, during therapy, and for six weeks after their last dose of EC MPS.

Exclusion Criteria:

1. Previous or planned kidney transplant.
2. Currently receiving continuous dialysis or GFR < 30 mL/min/1.73 m2 within 3 months prior to the start of study.
3. Patients with active serious digestive system disease, including infrequent cases of gastrointestinal tract ulceration with hemorrhage or perforation.
4. Patients currently with life threatening conditions including malignancies, or severe infection in recent 6 months prior to start of study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male and female patients diagnosed with LN between 20 and 75 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Safety profile of Enteric-coated Mycophenolate Sodium (EC-MPS) on Lupus nephritis patients | 12 months
  The primary endpoint is the safety of EC-MPS in LN patients, which will be assessed via the adverse events (AEs), serious adverse events (SAEs) and deaths.

SECONDARY OUTCOMES:
Reasons for study drug discontinuation | 12 months
  To describe the reasons for study drug discontinuation, including poor response, loss to follow-up, etc.
Proportion of patients with a complete response | month 6, month 12
  Patients will be reported to have a complete response if their proteinuria is < 0.5 g/24 hours; or UPCR≤ 0.5.
Proportion of patients with a partial response | month 6, month 12
  Patients will be reported to have a partial response if they experience any one criteria as follows:
  * At least 50% decrease from baseline in proteinuria. Note: patients with a baseline proteinuria of >3.5 g/24 hours, must have a proteinuria < 3 g/24 hours;
  * Red blood cells per high power field (RBCs/HPF) ≤50% above baseline and no RBC casts;
  * At least 50% decrease in UPCR or to <1.0 (if 1.0 ≤ baseline ≤3.0) or to ≤3.0 (if baseline was >3.0).
Proportion of patients achieving renal response in estimated glomerular filtration rate (eGFR) | month 6, month 12
  The proportion of patients achieving renal response in estimated glomerular filtration rate (eGFR).
  (eGFR within the normal range, or no less than 85% of baseline)
Proportion of patients achieving inactive urinary sediment | month 6, month 12
  The proportion of patients achieving inactive urinary sediment (no cellular casts)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Taiwan (5):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Keelung
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: No